CLINICAL TRIAL: NCT01828151
Title: Noninvasive Positive Airway Pressure Ventilation and Risk of Facial Pressure Ulcers in Patients With Acute Respiratory Failure
Brief Title: Noninvasive Positive Airway Pressure Ventilation and Risk of Facial Pressure Ulcers
Status: Completed | Type: Observational
Sponsor: Ospedale S. Giovanni Bosco (Other)
Responsible Party: Principal Investigator, Giovanni Ferrari, Dr, Ospedale S. Giovanni Bosco
Other Study IDs: gbosco5
Record Dates: First submitted 2013-03-21; First posted 2013-04-10 (Estimated); Last update posted 2013-04-10 (Estimated); Status verified 2013-04

CONDITIONS: Acute Respiratory Failure
Keywords: Pressure ulcer; Noninvasive ventilation
MeSH Terms: conditions — Pressure Ulcer

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Developed skin lesions: Patients treated with noninvasive ventilation for an episode of acute respiratory failure
  Interventions: Device: Noninvasive ventilation mask

INTERVENTIONS:
Device: Noninvasive ventilation mask
  Other Names: - Oro-nasal mask: Ultra Mirage NV, ResMed Australia; - Full-face mask: Performax, Respironics Inc USA; - Helmet: Castar R, StarMed - Mirandola Italy

SUMMARY:
To assess risk of skin pressure lesions in patients treated with noninvasive mechanical ventilation.

DETAILED DESCRIPTION:
Noninvasive ventilation improves the outcome of patients with acute respiratory failure; however patient's discomfort may be responsible for up to a fifth of failures. Scant literature exists on NIV-related pressure ulcers and their determinants.

Aim of the study is to seek for determinants, if any, associated with the development of pressure ulcers related to noninvasive ventilation.

Study design: observational. Patients treated with NIV from December 2009 to December 2011 will be analyzed. Main end-points: to seek for variables associated to the development of NIV-related pressure ulcers in patients with acute respiratory failure.

ELIGIBILITY:
Inclusion Criteria:

* severe dyspnea at rest
* respiratory rate > 30 per minute
* PaO2/FiO2 < 200 (despite oxygen with Venturi with a FiO2 og 0.5)
* use of accessory respiratory muscles
* pH < 7.35 > 7.10

Exclusion Criteria:

* STEMI
* NSTEMI/Unstable angina
* Hemodynamic instability
* Need for immediate endotracheal intubation
* Inability to protect the airways
* Impaired sensorium
* Pulmonary embolism
* Gastrointestinal bleeding
* Hematological malignancy or neoplasms with ECOG performance status > 2

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted to our high dependency unit for an episode of acute respiratory failure and treated with noninvasive ventilation.
Sampling Method: Non-Probability Sample
Enrollment: 170 (Actual)
Dates: Start 2009-12; Primary Completion 2011-12 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Risk of skin pressure ulcers in patients treated with noninvasive ventilation for acute respiratory failure. | Risk of pressure ulcers within 72 hours from noninvasive ventilation beginning.
  Skin lesions were classified as follows:
  * reddening,
  * loss of skin integrity,
  * necrotic lesion.

SECONDARY OUTCOMES:
Incidence of skin pressure ulcers in patients treated with noninvasive ventilation. | Incidence of skin pressure ulcers. Patients will be followed during duration of high dependency unit stay for an average length of stay of 7 days.
  Characterization of skin lesions during noninvasive ventilation in patients with acute respiratory failure.

CONTACTS AND LOCATIONS:
Overall Officials: Giovanni Ferrari, MD, Principal Investigator — Ospedale S. Giovanni Bosco
Locations (1):
- Medicina d'Urgenza - Terapia Subintensiva. Ospedale S. Giovanni Bosco, Torino, Torino, Italy